CLINICAL TRIAL: NCT05003934
Title: Safety of Cultured Allogeneic Adult Umbilical Cord Derived Mesenchymal Stem Cell Intravenous Infusion for the Treatment of Rheumatoid Arthritis
Brief Title: Safety of Cultured Allogeneic Adult Umbilical Cord Derived Mesenchymal Stem Cell Intravenous Infusion for RA
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The Foundation for Orthopaedics and Regenerative Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SC-8-ATG-10-03
Record Dates: First submitted 2021-08-06; First posted 2021-08-13 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment Group (Experimental): Single intravenous infusion of 100 million cells
  Interventions: Biological: AlloRx

INTERVENTIONS:
Biological: AlloRx — cultured allogeneic adult umbilical cord derived mesenchymal stem cells

SUMMARY:
This trial will study the safety and efficacy of intravenous infusion of cultured allogeneic adult umbilical cord derived mesenchymal stem cells for the treatment of Rheumatoid Arthritis

DETAILED DESCRIPTION:
Studies have shown that stem cell treatment is safe and efficacious for the treatment of Rheumatoid Arthritis (RA). Patients with RA will receive a single intravenous infusion of cultured allogeneic adult umbilical cord derived mesenchymal stem cells. The total dose will be 100 million cells. Patients will be evaluated within one month pre treatment and at 1, 6, 12, 24, 36, and 48 months post treatment for safety and efficacy.

For patients with more severe disease requiring chemotherapeutic drugs such as methotrexate, an autologous T Cell vaccine will be utilized created from the patient's own T cells obtained by apheresis

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Rheumatoid Arthritis
* Understanding and willingness to sign a written informed consent document

Exclusion Criteria:

* Active infection
* Active cancer
* Chronic multisystem organ failure
* Pregnancy
* Clinically significant Abnormalities on pre-treatment laboratory evaluation
* Medical condition that would (based on the opinion of the investigator) compromise patient's safety.
* Continued drug abuse
* Pre-menopausal women not using contraception
* Previous organ transplant
* Hypersensitivity to sulfur

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-11-07 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Safety (adverse events) | Four year follow-up
  Clinical monitoring of possible adverse events or complications

SECONDARY OUTCOMES:
Efficacy: the 28-joint disease activity score (DAS 28) | Four year follow-up
  DAS 28 is used to determine the disease activity for RA. It will be completed for each follow up point.
Efficacy: visual analog scale (VAS) | Four year follow-up
  VAS is a scale that is used to measure pain. It will be completed for each follow up point.

CONTACTS AND LOCATIONS:
Overall Officials: Chadwick Prodromos, MD, Principal Investigator — The Foundation for Orthopaedics and Regenerative Medicine
Locations (2):
- Medical Surgical Associates Center, St John's, Antigua and Barbuda
- Center for Investigation in Tissue Engineering and Cellular Therapy, Buenos Aires, Argentina

REFERENCES:
- [Background] Wells G, Becker JC, Teng J, Dougados M, Schiff M, Smolen J, Aletaha D, van Riel PL. Validation of the 28-joint Disease Activity Score (DAS28) and European League Against Rheumatism response criteria based on C-reactive protein against disease progression in patients with rheumatoid arthritis, and comparison with the DAS28 based on erythrocyte sedimentation rate. Ann Rheum Dis. 2009 Jun;68(6):954-60. doi: 10.1136/ard.2007.084459. Epub 2008 May 19. PMID 18490431
- [Background] Delgado DA, Lambert BS, Boutris N, McCulloch PC, Robbins AB, Moreno MR, Harris JD. Validation of Digital Visual Analog Scale Pain Scoring With a Traditional Paper-based Visual Analog Scale in Adults. J Am Acad Orthop Surg Glob Res Rev. 2018 Mar 23;2(3):e088. doi: 10.5435/JAAOSGlobal-D-17-00088. eCollection 2018 Mar. PMID 30211382
- [Background] Wang L, Huang S, Li S, Li M, Shi J, Bai W, Wang Q, Zheng L, Liu Y. Efficacy and Safety of Umbilical Cord Mesenchymal Stem Cell Therapy for Rheumatoid Arthritis Patients: A Prospective Phase I/II Study. Drug Des Devel Ther. 2019 Dec 19;13:4331-4340. doi: 10.2147/DDDT.S225613. eCollection 2019. PMID 31908418
- [Background] Ghoryani M, Shariati-Sarabi Z, Tavakkol-Afshari J, Ghasemi A, Poursamimi J, Mohammadi M. Amelioration of clinical symptoms of patients with refractory rheumatoid arthritis following treatment with autologous bone marrow-derived mesenchymal stem cells: A successful clinical trial in Iran. Biomed Pharmacother. 2019 Jan;109:1834-1840. doi: 10.1016/j.biopha.2018.11.056. Epub 2018 Nov 26. PMID 30551438